CLINICAL TRIAL: NCT07384338
Title: Three Dimensional Evaluation of Dento-Skeletal Effects of Leaf Self Expander in Cleft Lip and Palate Patients (A Randomized Controlled Clinical Trail)
Brief Title: Three Dimensional Evaluation of Dento-Skeletal Effects of Leaf Self Expander in Cleft Lip and Palate Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Tasneem Ahmed Almohamady Khalil, Assistant lecturer, Orthodontic Department, Faculty of Oral and Dental Medicine, MUST University., Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-OR-23-03
Record Dates: First submitted 2026-01-21; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Three Dimensional; Dento-Skeletal; Leaf Self Expander; Cleft Lip; Cleft Palate
MeSH Terms: conditions — Cleft Lip; Cleft Palate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Control group) (Active Comparator): Patients were treated with conventional therapy with rapid maxillary expansion (RME) for maxillary expansion.
  Patients were treated with Leaf Self Expander for maxillary expansion.
  Interventions: Other: Rapid maxillary expansion
- Group B (Tested group) (Experimental): Patients were treated with Leaf Self Expander for maxillary expansion.
  Interventions: Other: Leaf Self Expander

INTERVENTIONS:
Other: Rapid maxillary expansion — Patients were treated with conventional therapy with rapid maxillary expansion (RME) for maxillary expansion.
  Arms: Group A (Control group)
Other: Leaf Self Expander — Patients were treated with Leaf Self Expander for maxillary expansion.
  Arms: Group B (Tested group)

SUMMARY:
This study aims to evaluate the dento-alveolar changes after maxillary expansion in cleft lip and palate patients by Leaf Self Expander, as compared to conventional Rapid Maxillary Expander using digital cast analysis and three-dimensional cone-beam computed tomography.

DETAILED DESCRIPTION:
Orofacial clefts are the most prevalent among congenital malformations, which can involve the upper lip, alveolar ridge or/and the palate and, in general, cause esthetic, functional, and psychosocial impairments in different magnitudes, depending on its location and extension.

The Leaf Self Expander (LSE) is a new technology that similar to LE in design except absence of the reactivation screw and respects the principle of producing predetermined light, constant forces, without any intervention by the patient, parents or orthodontist. Where it is composed of three leaf springs compressed by the laboratory before delivery, it is deactivated spontaneously until the programmed expansion is achieved.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral or bilateral cleft lip and palate in mixed dentition.
* Lip and palate repair was performed from 3 to 24 months of age.
* Presence of maxillary constriction and need of maxillary expansion prior to secondary alveolar bone grafting.
* Good periodontal health.

Exclusion Criteria:

* Previous orthodontic treatments.
* Any systemic diseases.
* Multiple carious lesions.

Ages: 3 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Measurement of linear skeletal change | 6 months post-expansion
  Linear skeletal change was assessed to evaluate change in skeletal dimensions following the expansion procedure.

SECONDARY OUTCOMES:
Measurement of angular skeletal change | 6 months post-expansion
  Angular skeletal change was assessed to evaluate change in skeletal dimensions following the expansion procedure.
Measurement of linear dental change | 6 months post-expansion
  Linear dental change was assessed to evaluate change in tooth position and arch dimensions following the expansion procedure.
Measurement of angular dental change | 6 months post-expansion
  Angular dental change was assessed to evaluate change in tooth position and arch dimensions following the expansion procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.